CLINICAL TRIAL: NCT02931422
Title: Financial Incentives to Increase Pediatric HIV Testing Pilot Study
Brief Title: Financial Incentives to Increase Pediatric HIV Testing Pilot Study (FIT-Pilot)
Acronym: FIT-Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Kenyatta National Hospital (Other Government); University of Nairobi (Other)
Responsible Party: Principal Investigator, Jennifer Slyker, Assistant Professor, Global Health, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 50526-J
Record Dates: First submitted 2016-10-07; First posted 2016-10-13 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-02

CONDITIONS: HIV
Keywords: HIV; financial incentive; pediatric HIV testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low Financial Incentive (Experimental): Conditional cash transfer upon HIV testing
  Interventions: Behavioral: Financial incentive
- Medium Financial Incentive (Experimental): Conditional cash transfer upon HIV testing
  Interventions: Behavioral: Financial incentive
- High Financial Incentive (Experimental): Conditional cash transfer upon HIV testing
  Interventions: Behavioral: Financial incentive

INTERVENTIONS:
Behavioral: Financial incentive — Conditional cash transfer upon HIV testing

SUMMARY:
The aim of the pilot study is to evaluate the feasibility, acceptability and costs of a financial incentive intervention to motivate pediatric HIV testing in Western Kenya. The study will evaluate 3 cash incentive values and determine percent uptake of testing. A post-test questionnaire will explore parental satisfaction, mechanisms of incentive effectiveness and the impact of testing on emotional health and pediatric healthcare utilization.

DETAILED DESCRIPTION:
The study will be a randomized trial with 3 arms (1:1:1 allocation) with small, medium, and large cash incentive. The investigators will randomize 60 parents with children of unknown status at Kisumu County Hospital in Western Kenya.

ELIGIBILITY:
Inclusion Criteria:

* Parent/caregiver receiving HIV care
* Parent/caregiver is female
* Parent/caregiver has one or more children <13 years old
* Child is HIV exposed (parent/caregiver report or clinic confirmation)
* Caregiver reports child's HIV status is unknown

Exclusion Criteria:

-None

*The investigators reserve the right to exclude any potential enrollee who is deemed to be a high personal risk, or whose children are at high personal risk, of interpersonal violence, by study participation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-01-31 (Actual); Study Completion 2017-01-31 (Actual)

PRIMARY OUTCOMES:
HIV testing | Testing within 2 months of recruitment
  % of parents completing pediatric HIV testing within 2 months will be compared between arms.

SECONDARY OUTCOMES:
Parental satisfaction with incentives | 2 months of recruitment
  A post-test questionnaire will assess parental satisfaction with the incentive, including the value provided, other preferred formats (vouchers, agricultural items, etc)
Motivational mechanism | 2 months
  A post-test questionnaire will assess mechanisms by which incentives motivate behavioral change. Questions will assess potential for coercion, parental previous intention to test, and whether incentives overcame economic and/or emotional barriers to testing
Care seeking | 2 months
  A post-test questionnaire will assess whether learning the child's HIV status will affect the likelihood of seeking future medical services for the child
Emotional impact | 2 months
  A post-test questionnaire will assess impact of testing on caregiver, child, and family emotional well-being

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer A Slyker, PhD, MSc, Principal Investigator — University of Washington; Irene N Njuguna, MBChB, Msc, Principal Investigator — University of Washington/Kenyatta National Hospital
Locations (1):
- Kisumu County Hospital, Kisumu, Kenya